CLINICAL TRIAL: NCT01007838
Title: Effects of Progressive Resistance Training During Haemodialysis on Muscle Quantity and Function in Patients With Chronic Kidney Disease
Brief Title: Intradialytic Progressive Resistance Training for Maintenance Haemodialysis Patients
Acronym: PRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangor University (Other)
Collaborators: Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R& D Ref no: MACDONALD 07/53
Record Dates: First submitted 2009-10-15; First posted 2009-11-04 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Kidney Disease
Keywords: Progressive Resistance Training/Exercise; Muscle wasting; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chronic kidney disease progressive resistance training group (Experimental): Progressive resistance training programme using a dialysis specific fitness machine: 80 % of predicted one repetition max, weight lifted will be increased when three sets of ten repetitions can be completed without failure.
  Interventions: Other: Progressive resistance training programme
- Chronic kidney disease sham exercise group (Sham Comparator): Lower body stretching exercise using the easiest rehabilitation elastic Theraband
  Interventions: Other: Sham exercise
- Healthy controls progressive resistance training group (Experimental): Progressive resistance training programme using a dialysis specific fitness machine: 80 % of predicted one repetition max, weight lifted will be increased when three sets of ten repetitions can be completed without failure.
  Interventions: Other: Progressive resistance training
- Healthy controls sham exercise group (Sham Comparator): Lower body stretching exercise using the easiest rehabilitation elastic Theraband
  Interventions: Other: Sham exercise

INTERVENTIONS:
Other: Progressive resistance training programme — Progressive resistance training programme using a dialysis specific fitness machine: 80 % of predicted one repetition max, weight lifted will be increased when three sets of ten repetitions can be completed without failure.
  Other Names: Intradialytic resistance exercise
  Arms: Chronic kidney disease progressive resistance training group
Other: Sham exercise — Lower body stretching exercise using the easiest rehabilitation elastic Theraband
  Arms: Chronic kidney disease sham exercise group
Other: Progressive resistance training — Progressive resistance training programme using a dialysis specific fitness machine: 80 % of predicted one repetition max, weight lifted will be increased when three sets of ten repetitions can be completed without failure.
  Arms: Healthy controls progressive resistance training group
Other: Sham exercise — Lower body stretching exercise using the easiest rehabilitation elastic Theraband
  Arms: Healthy controls sham exercise group

SUMMARY:
The purpose of this study is to investigate the effects of a 12 week progressive resistance training during haemodialysis on muscle quantity and physical functioning in chronic kidney disease patients receiving maintenance haemodialysis.

It is hypothesised, based on previous literature involving similar resistance training protocols in other catabolic conditions, that the resistance training will result in a significant increase in muscle quantity as well a physical function.

DETAILED DESCRIPTION:
Muscle wasting is common in patients with chronic kidney disease and has been associated with decreased ability to complete activities of daily living, increased hospitalisation and therefore and decreased quality of life.

In other catabolic conditions, such as cancer or rheumatoid arthritis, exercise is an established treatment to reverse muscle wasting. It is uncertain whether exercise has this effect in the chronic kidney disease population due to an altered hormone system that may prevent the anabolic effects of exercise from occurring. However, progressive resistance training, which is exercise that is most effective at eliciting an anabolic response has not been effectively carried out with haemodialysis patients.

Therefore, this study aims to investigate whether or not a twelve week intradialytic progressive resistance training programme will have an effect on muscle quantity, physical function and quality of life in patients receiving maintenance haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney diseases stage five requiring maintenance hemodialysis.

Exclusion Criteria:

* Patients who have been receiving dialysis for less than 3 months;
* Are under the age of 18years;
* Have medical contradictions to participate in the exercise programs;
* Any uncontrolled medical condition which does not allow participation in exercise;
* Have known neuro-muscular disorders;
* Have any other uncontrolled medical condition, including pregnancy;
* Are not independently ambulant for 50 m;
* Have received anabolic intervention, or had catabolic conditions within the last 3 months;
* Have a cardiac pacemaker or other unsuitable implanted device for magnetic resonance;
* Are vulnerable to heat stress;
* Or are unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie H MacDonald, PhD, Principal Investigator — Bangor University
Locations (1):
- Renal unit, Ysbyty Gwynedd, North West Wales NHS Trust, Bangor, Gwynedd, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronic kidney patients were recruited from local renal units. Healthy controls were recruited from the North Wales Community. Recruitment period was from January 2009 to July 2011.
Period: Overall Study
Arm/Group | Chronic Kidney Disease Progressive Resistance Training Group | Chronic Kidney Disease Sham Exercise Group | Healthy Controls Progressive Resistance Training Group | Healthy Controls Sham Exercise Group
Started | 12 | 11 | 5 | 4
Completed | 9 | 11 | 5 | 4
Not Completed | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Started home haemodialysis | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease Progressive Resistance Training Group | Chronic Kidney Disease Sham Exercise Group | Healthy Controls Progressive Resistance Training Group | Healthy Controls Sham Exercise Group | Total
Number analyzed (Participants) | 12 | 11 | 5 | 4 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 4 | 4 | 22
  >=65 years | 4 | 5 | 1 | 0 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (18) | 67 (16) | 51 (13) | 40 (17) | 51 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 4 | 16
  Male | 7 | 7 | 2 | 0 | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 11 | 5 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Muscle Cross Sectional Area
Description: Muscle cross sectional area (quadriceps group) taken at midpoint slice between superior aspect of femoral head and the femoral condyle.
Time Frame: Change from baseline in cross sectional area at 12 weeks
Population: Per protocol. All participants completing the study were analyzed.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Chronic Kidney Disease Progressive Resistance Training Group | Chronic Kidney Disease Sham Exercise Group | Healthy Controls Progressive Resistance Training Group | Healthy Controls Sham Exercise Group
Number analyzed (Participants) | 9 | 11 | 5 | 4
cm2 | 3.24 (5.10) | -4.62 (6.33) | 4.39 (3.43) | -0.15 (2.10)
Statistical Analysis 1: Comparison: Chronic Kidney Disease Progressive Resistance Training Group vs Chronic Kidney Disease Sham Exercise Group vs Healthy Controls Progressive Resistance Training Group vs Healthy Controls Sham Exercise Group; Omnibus ANCOVA. An interaction would suggests patients responded to exercise differently than controls; Test type: Superiority or Other; p = 0.30, ANCOVA — Statistical significance was accepted if p < 0.05
Statistical Analysis 2: Comparison: Chronic Kidney Disease Progressive Resistance Training Group vs Chronic Kidney Disease Sham Exercise Group; Follow up ANOVA in chronic kideny disease patients only. An interaction would suggest patients allocated to the resistance exercise group increased muscle size more than those allocated to the sham exercise group; Test type: Superiority or Other; p = 0.0017, ANOVA — Statistical significance was accepted if p < 0.05
Statistical Analysis 3: Comparison: Healthy Controls Progressive Resistance Training Group vs Healthy Controls Sham Exercise Group; Follow up ANOVA in healthy controls only. An interaction would suggest healthy controls allocated to the resistance exercise group increased muscle size more than those allocated to the sham exercise group; Test type: Superiority or Other; p = 0.024, ANOVA — Statistical sigficance was accepted if p < 0.05

2. Secondary Outcome: Muscle Strength
Description: Bilateral knee extensor isometric strength.
Time Frame: Change from baseline in muscle strength at 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Chronic Kidney Disease Progressive Resistance Training Group | Chronic Kidney Disease Sham Exercise Group | Healthy Controls Progressive Resistance Training Group | Healthy Controls Sham Exercise Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
Small sample size in healthy control group. Variable gender mix in all groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes